CLINICAL TRIAL: NCT04276389
Title: OCT- Versus Angiography-guided Paclitaxel Drug-Coated Balloon Angioplasty in De Novo Coronary Artery After Lesion Preparation With Scoring Balloon - A Prospective Multicenter Cohort Study
Brief Title: OCT- Versus Angiography-guided Paclitaxel Drug-Coated Balloon Angioplasty in De Novo Coronary Artery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018015
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided arm (Active Comparator)
  Interventions: Device: OCT-guided paclitaxel drug-coated balloon angioplasty
- Angiography-guided arm (Placebo Comparator)
  Interventions: Device: Angiography-guided paclitaxel drug-coated balloon angioplasty

INTERVENTIONS:
Device: OCT-guided paclitaxel drug-coated balloon angioplasty — OCT-guided paclitaxel drug-coated balloon angioplasty in middle-sized de novo coronary artery
  Arms: OCT-guided arm
Device: Angiography-guided paclitaxel drug-coated balloon angioplasty — Angiography-guided paclitaxel drug-coated balloon angioplasty in middle-sized de novo coronary artery
  Arms: Angiography-guided arm

SUMMARY:
OCT allows precise evaluation of intimal injury after lesion preparation and may improve the acute results and long-term outcomes after paclitaxel drug-coated balloon angioplasty. This prospective multicenter cohort study aims to assess the efficacy and safety of OCT- versus angiography-guided paclitaxel drug-coated balloon angioplasty in middle-sized de novo coronary artery after lesion preparation with scoring balloon.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years old
2. Patients have ischemic symptoms or evidence of myocardial ischemia (inducible or spontaneous) in the presence of a stenosis of at least 50% in a native coronary artery, including stable angina, unstable angina, or silent ischemia.
3. Reference vessel diameter >2.5 mm, and <4.0 mm.
4. Lesion length of <22 mm
5. Written informed consent

Exclusion Criteria:

1. Myocardial infarction within 4 weeks, including ST-elevation myocardial infarction and non-ST-elevation myocardial infarction
2. Cardiogenic shock (systolic arterial pressure <90mmHg), congestive heart failure (NYHA or Killip≥3)
3. Chronic kidney disease (eGFR <30 ml/min)
4. Lesion length >22 mm, or vessel diameters of <2.5 mm or >4.0 mm
5. Stents covering a major side branch (>2 mm)
6. Left main lesion
7. Graft lesion
8. Aortic-coronary ostial lesion
9. In-stent restenotic lesion
10. Chronic total occlusion
11. Severe calcified lesions.
12. Visible angiographic thrombus
13. Severe comorbidities: eg. malignancy (life expectancy <2 years)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss | 9 months
  Evaluated by QCA

SECONDARY OUTCOMES:
Rate of binary restenosis | 9 months
  Evaluated by QCA
Target lesion failure | 9 months
  Including death, target vessel myocardial infarction, or target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided